CLINICAL TRIAL: NCT04636645
Title: Effects of Lower Limb Positive Pressure on the Balance of Community-dwelling Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/0011961
Record Dates: First submitted 2020-11-08; First posted 2020-11-19 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Old Age; Fall

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Treadmill (Active Comparator): After completion of the baseline evaluation, Group A participants will exercise for 25 minutes under low-load walking conditions three times a week for 8 consecutive weeks on the AGT treadmill at a set speed of 3.1 mph at a 0-degree incline. For each session, 20% support will be given to participants
  Interventions: Other: Normal treadmill
- Anti-gravity treadmill with lower limb positive pressure (Experimental): Group B participants will be exercised for 25 minutes under normal-load walking conditions three times a week for 8 consecutive weeks on the AGT treadmill at a set speed of 3.1 mph at a 0-degree incline. Participants will be blinded to the study groups.
  Interventions: Other: Anti-gravity treadmill with lower limb positive pressure
- Anti-gravity treadmill with without lower limb positive pressure (Experimental): Group C participants will be exercised for 25 minutes three times a week for 8 consecutive weeks on the normal treadmill at a set speed of 3.1 mph at a 0-degree incline. Participants will be blinded to the study groups.
  Interventions: Other: Anti-gravity treadmill with without lower limb positive pressure

INTERVENTIONS:
Other: Normal treadmill — Participants will exercise for 25 minutes under low-load walking conditions three times a week for 8 consecutive weeks on the AGT treadmill at a set speed of 3.1 mph at 0-degree incline. For each session, 20% support will be given to participants.
  Arms: Normal Treadmill
Other: Anti-gravity treadmill with lower limb positive pressure — Participants will be exercised for 25 minutes under normal-load walking conditions three times a week for 8 consecutive weeks on the AGT treadmill at a set speed of 3.1 mph at 0-degree incline. Participants will be blinded to the study groups.
  Arms: Anti-gravity treadmill with lower limb positive pressure
Other: Anti-gravity treadmill with without lower limb positive pressure — Participants will be exercised for 25 minutes three times a week for 8 consecutive weeks on the normal treadmill at a set speed of 3.1 mph at a 0-degree incline. Participants will be blinded to the study groups.
  Arms: Anti-gravity treadmill with without lower limb positive pressure

SUMMARY:
With the onset of the sixth decade in life, degenerative processes affect the neuromuscular system in terms of losses in muscle strength (dynapenia) and muscle mass (sarcopenia). Neural (e.g., numerical loss of alpha motoneurons) and morphological factors. Borde et al. 123 number and size of particularly type-II muscle fibers), as well as their interaction, are responsible for age-related declines in muscle strength and mass. There is evidence that muscular weakness is highly associated with impaired mobility and an increased risk for falls. Moreover, lower extremity muscle weakness was identified as the dominant intrinsic fall-risk factor with a five-fold increase in the risk of falling. An anti-gravity treadmill allows users to walk or run in a reduced body weight environment. The user walks or runs on a treadmill belt surrounded by an enclosed, air-filled chamber. When air pressure increases, an upward force offloads the weight of the runner and decreases the percentage of body weight (BW%) experienced upon foot impact. So, a research question was developed in our mind after the literature review. Is there any effect of AGT training on fall risk of older adults?

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling adults aged 55 years and above.
2. Berg balance score should be from 46 to 54.
3. Able to follow instructions in Urdu.
4. No neurological conditions, and no musculoskeletal injuries within the past year.
5. Both male and female.

Exclusion Criteria:

1. Pain with ambulation or dizziness when standing or walking.
2. Contraindications to treadmill walking and LBPP such as cardiovascular conditions.
3. Severe osteoporosis, fractures, when loading of the abdominal region, hip or pelvis is contraindicated (such as groin infections, skin graft in the groin region, gastrointestinal tubes, colostomy, compromised skin integrity), orthopedic conditions in the past year or neurological conditions.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | 12 week
  Test is also commonly used to evaluate fall risk.A faster time for completion of required task indicates a better ability to perform functional activities. The person sits up from the chair after instruction and walks at his normal pace for 3 meters, takes a turn and sits down after walking back towards the chair. The total duration required for this activity is measured using a stop watch.
Berg balance scale | 12 week
  Evaluation of functional balance was done using BBS which is valid and reliable tool for dynamic and static balance assessment. It consists of 14 Items and balance is assessed using an ordinal scale comprising 5 points that ranges from 0 to 4. High scores are indicative of superior balance where as low scores are suggestive of increased fall risk and poor balance.
Functional reach test | 12 week
  This test is used to assess stability level of patient. The assessment is carried out by calculating the maximum distance a person is able to reach forward in a fixed standing position. The assessment is carried out by calculating the maximum distance a person is able to reach forward in a fixed standing position. Lower distance of functional reach test indicated higher risk of fall and deteriorated balance and vice versa.
Fall risk score | 12 week
  FRS provide an objective assessment of static and dynamic balance and was assessed using dynamic posturo graphy system. High scores of FRS indicated higher risk of fall and deteriorated balance and vice versa.
Balance App | 12 week
  There are six different tasks that subject have perform with system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and close and standing on a compromised surface with eyes open and close. High scores indicated higher risk of fall and deteriorated balance and vice versa.

SECONDARY OUTCOMES:
Force Plate | 12 week.
  Force plates is portable, non-invasive and quantitative instrument used to measure the ground reaction forces, variation in center of gravity and forces impact on foot. Postural sways will be calculated from force plate data. Randomness in data show increase risk of fall and poor balance.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No